CLINICAL TRIAL: NCT01819792
Title: Incidence of Respiratory Viral Infections During AML Induction and Consolidation Chemotherapy
Brief Title: Respiratory Viral Infections During Acute Myeloid Leukemia (AML)Chemotherapy Related Aplasia
Acronym: LAMVIRE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2011_843_0005
Record Dates: First submitted 2013-03-18; First posted 2013-03-28 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patient with Acute Myeloïd Leukemia (Other)
  Interventions: Other: Multiplex respiratory viral PCR

INTERVENTIONS:
Other: Multiplex respiratory viral PCR

SUMMARY:
Infectious morbidity and mortality is a major complication of AML (Acute Myeloid Leukemia) induction and consolidation chemotherapies related aplasia. The main aim of this study is to measure incidence of respiratory viral infections during AML induction and consolidation chemotherapy related aplasia. Primary end point is a positive polymerase chain reaction(PCR)associated with clinical signs.

DETAILED DESCRIPTION:
Bacterial and fungal infection treatment is well defined with guidelines. Few data are available for viral infections and concern essentially allogeneic stem cell transplantation. These infections are associated with a high mortality and morbidity rate. Data concerning AML are essentially retrospective, pediatric and with a little number of patients. Respiratory viral infections incidence is not known. These infections may be responsible for a higher mortality rate. Different risk factors are found: age superior to 65 years, lymphopenia, co-infections. Treatment is subject to a controversy: surveillance or starting an antiviral therapy. This study aims at understanding viral infections epidemiology during long term aplasia and optimizing their management.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old with an AML diagnostic and treated with induction and consolidation chemotherapy. Patients enrolled in another protocol may be included.
* Patients with relapsed leukemia who are treated with a salvage intensive therapy stay in the study
* Patients who have signed a consent policyholder

Exclusion Criteria:

* patients under 18 years old
* patients treated with another treatment than induction and consolidation chemotherapy
* pregnant women
* patients HIV, HBV or HBC positive
* patients with a positive PCR at J1
* patients treated with an antiviral treatment or an immunosuppressive treatment for another pathology
* patients under guardianship
* Primitive immunity Deficit

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2013-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
positivity of the viral PCR in the presence of clinical signs during periods of positivity of the PCR in the presence of clinical signs | at day 15
  Positivity of the viral PCR in the presence of clinical signs during periods of Aplasia following chemotherapy induction and consolidation defining viral infection.

SECONDARY OUTCOMES:
seasonal viral infection incidence measure | 18 months after inclusion
risk factor of viral infections research | 18 months after inclusion
viral infections related morbidity and mortality estimation | 18 months after inclusion
bacterial and fungal co-infection estimation | 18 months after inclusion
description of antiviral therapeutic used for treating patients | 18 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Jean Pierre MAROLLEAU, MD PHD, Principal Investigator — CHU AMIENS; FABRICE JARDIN, MD PHD, Principal Investigator — CHU ROUEN; OUMEDALY RENAN, MD PHD, Principal Investigator — CHU CAEN; BRUNO QUESNEL, MD PHD, Principal Investigator — CHRU LILLE
Locations (4):
- France (4):
  - Pr Marolleau, Amiens
  - CHU CAEN, Caen
  - Chru Lille, Lille
  - Chu Rouen, Rouen